CLINICAL TRIAL: NCT05713084
Title: Assessment of Condylar Position Changes and TMJ Functions After BSSO Mandibular Setback, Low Medial vs High Medial Cut (Randomized Controlled Trial)
Brief Title: Condylar Position Changes and TMJ Functions After BSSO Mandibular Setback, Low Medial Cut.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohammed Mahmoud Hussein Alaswad, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14922
Record Dates: First submitted 2023-01-21; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Maxillofacial Abnormalities; Mandible Prognathism; Skeletal Malocclusion
Keywords: mandibular setback; low medial cut; condylar position
MeSH Terms: conditions — Maxillofacial Abnormalities; Malocclusion, Angle Class III

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mandibular setback using low medial cut ostetomy (Experimental): mandibular setback using low medial cut ostetomy by keeping the cut ''low'' or close to the mandibular occlusal plane and ''short'' or terminating anterior to the lingula.
  Interventions: Other: mandibular setback using BSSRO
- mandibular setback using high medial cut ostetomy (Active Comparator): mandibular setback by placement of the medial ramus osteotomy cut 'high', just a few millimeters above the lingula, superior and lateral to the entrance point of the inferior alveolar nerve (IAN) into the mandibular foramen ,
  Interventions: Other: mandibular setback using BSSRO

INTERVENTIONS:
Other: mandibular setback using BSSRO — mandibular setback using BSSRO

SUMMARY:
This study hypotheses that using low medial cut osteotomy BSSO in mandibular setback can be an efficient and effective method to limit the bony segment interferences , decreasing muscles stripping during osteotomy ,decrease condylar torque and so securing preoperative condylar position during BSSO in comparison with using high medial cut BSSO.

DETAILED DESCRIPTION:
Research question:

Description of research question:

P: Population: Patients with facial skeletal deformity and need for mandibular setback using bilateral sagittal split osteotomy (BSSRO) alone or combined with lefort osteotomy.

I: Intervention: Patients with facial skeletal deformity and need and for mandibular setback using low medial cut osteotomy as modification of bilateral sagittal split ramus osteotomy (BSSRO).

C: Comparator: Patients with facial skeletal deformity and need and for mandibular setback using traditional high medial cut osteotomy bilateral sagittal split ramus osteotomy (BSSRO).

O: Outcome: Comparing the post-operative condylar positions changes and TMJ functions of two osteotomies.

Research question:

Is using low medial cut osteotomy modification in BSSRO in mandibular setback will provide more control over proximal segment position than traditional high medial cut through:

1. limit the segments interference and so maximizes the passive bony contact across the osteotomy site after surgically repositioning the distal segment
2. Passively positioned the proximal segment without displacement of the condyle from its normal position.

ELIGIBILITY:
Inclusion criteria:

* Age of the patient between (18-60) years
* Patients in need of mandibular setback using bilateral sagittal split osteotomy.
* All patients are free from any systemic disease that may affect normal bone healing.
* Patient with facial deformity will be treated with mandibular setback either mono or bimaxilary surgeries
* Patient with facial deformity will be treated with mandibular setback either surgery first approach or orthofirst approach.
* Sufficient dentition to reproduce the occlusal relationships
* Patient's consent to participate

Exclusion criteria:

* Patients with any systemic disease that may affect normal healing
* Intra-bony lesions or infections that may interfere with surgery.
* Previous orthognathic surgeries.
* Patients with all types of facial clefts

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
3D mandibular condylar position changes | Preoperative- 1-month postoperative - 6 months post operative
  assessment of condylar position changes in millimetre using C.T.(axial ,coronal and sagital cut. ).
  1. Axial condylar head long-axis angle (AHA):
     angle between the sagittal plane and the axial condylar head axis line
  2. Axial condylar head position (AHP):
     perpendicular distance between the sagittal plane and the most medial point of the condylar head
  3. Frontal condylar head long-axis angle (FHA):
     angle between the axial plane and the frontal condylar head long-axis line
  4. Frontal condylar head position (FHP):
     perpendicular distance between the axial plane and most superior point of the condylar head
  5. Sagittal condylar head long-axis angle (SHA):
     angle between the coronal plane and the sagittal condylar head long-axis line
  6. Sagital condylar head position (SHP):
  perpendicular distance between the coronal plane and the most superior point of the condylar head

SECONDARY OUTCOMES:
Assessment of changes in articular disc position | Preoperative , 6month postoperative
  In order to trace the position of the TMJ disc, a line was drawn from the uppermost point of the articular fossa (UAF, marked as 10) to the lowermost point of the articular tubercle (LAT, marked as 0).
  This line was continued anteriorly and inferiorly. If the anterior border of the disc was anterior to this line, it was considered negative. These two points were chosen because they did not change with remodelling .
  Perpendicular lines to this line were drawn in the anterior and posterior borders of the disc. Finally, disc position was determined by averaging anterior (point A) and posterior (point P) disc limits.

OTHER OUTCOMES:
Clinical assessment of maximum incisal opening (MIO) | Preoperative - 1 months postoperative - 6 months postoperative
  assessment of changes(in millimetre) in Maximum incisal opening (MIO)
pain on TMJ | Preoperative - 1 months postoperative - 6 months postoperative
  assessment of changes in severity of pain over TMJ using (pain scale from 0 to 10)
sounds on TMJ | Preoperative - 1 months postoperative - 6 months postoperative
  assessment of resulted sounds during TMJ function (present or not present)

CONTACTS AND LOCATIONS:
Overall Officials: Fahmy Mobarak, professor, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt